CLINICAL TRIAL: NCT07337434
Title: Comparison of Efficacy of Methotrexate vs Apremilast in Moderate to Severe Plaque Psoriasis
Brief Title: To Check Comparison of Apremilast and Methotrexate Efficacy in Patients With Moderate to Severe Plaque Psoriasis Presented to Tertiary Care Hospital
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Syeda Sana Zaman (Other Government)
Responsible Party: Sponsor-Investigator, Syeda Sana Zaman, Training medical officer, Hayat Abad Medical Complex, Peshawar
Organization: Hayat Abad Medical Complex, Peshawar (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HayatabadMC
Record Dates: First submitted 2025-12-17; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Chronic Plaque Psoriasis
MeSH Terms: interventions — Methotrexate; apremilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methotrexate (Experimental): This group will recieve methotrexate 10-25mg once weekly for 3 months,
  Interventions: Drug: Methotrexate
- Apremilast (Experimental): This group will recieve apremilast 30mg BD for 3 months.
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Methotrexate — Group A will recieve methotrexate 10-25mg once weekly for 3 months. Along with folic acid once daily except on day of methotrexate.
  Arms: Methotrexate
Drug: Apremilast — Group B will recieve tablet apremilast 30mg twice daily for 3 months.
  Arms: Apremilast

SUMMARY:
This study aims to compare efficacy of methotrexate vs apremilast in the management of chronic plaque psoriasis.Given the high prevalence of psoriasis in Pakistan and the significant psychological impact on patients, particularly in Peshawer,this study will provide valuable insights into optimal treatment strategies.

DETAILED DESCRIPTION:
Introduction Plaque Psoriasis are red, scaly plaques which mostly manifests on the skin's extensor surfaces, are the hallmark of plaque psoriasis, a chronic inflammatory skin disorder. It significantly impairs patients' quality of life and poses therapeutic challenges due to chronicity and relapse tendency. Approximately 2% to 3% of the global population deals with psoriasis. The most frequent subtype of psoriasis, plaque psoriasis, affects between 0.5% to 1% of Pakistanis, according to research conducted in hospitals.

Patients with moderate to severe disease were traditionally treated with methotrexate-based systemic therapy. However, its long-term safety profile concerning hepatotoxicity and myelosuppression requires periodic monitoring. Apremilast, a newer oral phosphodiesterase-4 inhibitor, has demonstrated moderate efficacy with a favorable safety profile but is less commonly used in developing countries due to cost and limited availability.

While multiple studies have evaluated the efficacy of both drugs individually, direct head-to-head comparisons in regional populations are lacking. Recent international trials indicate Apremilast may have a better tolerability profile but lower efficacy compared to Methotrexate.Apremilast was reported to be more effective than methotrexate (47.3% vs 21.8%) in decreasing PASI scores over 12 weeks in a recent research involving 112 individuals with moderate to severe plaque psoriasis. Both therapies had minor adverse effects, but Apremilast was found to be more effective.

Despite methotrexate's extensive use in treating moderate to severe plaque psoriasis, concerns regarding its long-term safety and variable effectiveness persist. Apremilast, a newer oral agent, offers a favorable safety profile but is underutilized in resource-limited settings due to cost and limited availability. Few local studies have compared the two treatments using PASI and other standardized outcome measures to determine whether one is more effective. In light of the relative efficacy and safety of Methotrexate and Apremilast, it is imperative that Pakistani physicians have access to the findings of this trial so that they may make treatment decisions grounded in data.

Objective To compare the efficacy of methotrexate vs apremilast in moderate to severe plaque psoriasis.

Operational Definitions

Moderate to Severe Plaque Psoriasis:

Moderate to severe disease will be defined as PASI ≥10. Diagnosis will be confirmed by consultant dermatologist using clinical criteria and PASI tool. (Annex-A)

Efficacy:

Efficacy will be assessed based on reduction in PASI score from baseline to 12 weeks. A 75% reduction in PASI score from the baseline will be considered as primary efficacy outcome.

Null Hypothesis (H₀): When it comes to treating moderate to severe plaque psoriasis, there is statistically insignificant difference between Apremilast and Methotrexate.

Alternate Hypothesis (H₁): In terms of reducing PASI scores, Apremilast is statistically superior to Methotrexate for treating moderate to severe plaque psoriasis.

Material and Methods

Study Design:

Randomized Control Trial

Study Setting:

Department of Dermatology, MTI-Hayatabad Medical Complex (HMC), Peshawar

Duration of Study:

Six months after approval.

Sample Size: Using WHO sample size calculator, with anticipated efficacy of Methotrexate as 21.80% and Apremilast as 47.3%⁹, 95% confidence level, 80% power, the calculated sample size is 106 patients (53 in each group).

Sampling Technique:

Random Sampling

Inclusion Criteria:

Patients having age between 18-60 years of either gender Diagnosed with moderate to severe plaque psoriasis (PASI ≥10) No prior systemic therapy in past 3 months.

Exclusion Criteria:

Pregnancy or lactation History of liver or renal dysfunction Known hypersensitivity to study drugs

Data Collection Procedure This study will be conducted at the Department of Dermatology, MTI-Hayatabad Medical Complex, Peshawar, following formal approval from the Hospital Ethical Committee and CPSP Karachi. Random sampling will be used to recruit patients who fulfill the inclusion criteria and give written informed consent. When PASI scores (Annex-A) indicate moderate to severe plaque psoriasis, a consulting dermatologist will confirm the diagnosis. After a comprehensive clinical evaluation of each participant using block randomization, eligible patients will be divided into two therapy groups: Group A, which will get 10-25 mg of methotrexate once weekly along with folic acid supplements, and Group B, which will receive 30 mg of Apremilast twice daily following dose titration. Baseline PASI scores and demographic data will be recorded on a structured data collection form. Follow-up evaluations will be scheduled at the 4th, 8th, and 12th week of therapy to assess treatment efficacy, monitor for adverse effects, and ensure compliance. PASI scoring will be repeated at each visit, and any side effects or treatment modifications will be documented accordingly. Using a pre-made proforma, all data will be recorded.

Data Analysis Procedure:

The Statistical Package for the Social Sciences, version 26.0, will be used to input and analyze the data. Age and PASI score will be examined using the Shapiro-Wilk test to check normality. Mean+SD/Median (IQR) will be used for numerical variables. Categorical variables, such as gender, treatment group, demographics and efficacy, will be summarized using frequencies and percentages. An independent samples t-test will be conducted to evaluate the treatment efficacy of the Apremilast and Methotrexate groups based on the mean reduction in PASI scores. To compare categorical variables with efficacy, a chi-square test or Fisher's exact test will be utilized, with a p value less than 0.05 being considered statistically .

ELIGIBILITY:
Inclusion Criteria:

Patients having age between 18-60 years of either gender Diagnosed with moderate to severe plaque psoriasis (PASI ≥10) No prior systemic therapy in past 3 months.

Exclusion Criteria:

Pregnancy or lactation History of liver or renal dysfunction Known hypersensitivity to study drugs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2026-06-25 (Estimated); Study Completion 2026-06-25 (Estimated)

PRIMARY OUTCOMES:
PASI SCORE calculation | 3 months
  Efficacy of drugs are measured by calculation of PASI score for both groups at each visit.A treatment will be deemed effective if it achieves 75% reduction in PASI score from the baseline in 12 weeks.
  Score ranges from 0 (no disease) to 72( maximums severity)
  Interpretation:
  0-5 mild 6-10 moderate >10 severe

CONTACTS AND LOCATIONS:
Locations (1):
- MTI-HMC Peshawar, Peshawar, Khyber Pukhtunkhwa, Pakistan